CLINICAL TRIAL: NCT01128972
Title: Evaluation of a Test Mouthwash and Dentifrice Regimen in an In-situ Model of Dental Erosion
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: Z3480664
Record Dates: First submitted 2010-04-30; First posted 2010-05-24 (Estimated); Results first posted 2013-04-25 (Estimated); Last update posted 2015-01-01 (Estimated); Status verified 2014-12

CONDITIONS: Tooth Erosion
Keywords: enamel erosion; tooth remineralization; tooth erosion
MeSH Terms: conditions — Tooth Erosion | interventions — Sodium Fluoride

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (5):
- Test Dentifrice + Test Mouth Rinse (MR) (Experimental): Test fluoride dentifrice and test fluoride MR
  Interventions: Drug: Sodium fluoride
- Test Dentifrice + Sterile Water Rinse (Experimental): Test fluoride dentifrice and sterile water rinse
  Interventions: Drug: Sodium fluoride; Drug: Sterile water
- Placebo Dentifrice + Test MR (Experimental): Placebo dentifrice and test fluoride rinse
  Interventions: Drug: Sodium fluoride
- Reference Dentifrice + Sterile Water Rinse (Active Comparator): Marketed fluoride dentifrice with sterile water rinse
  Interventions: Drug: Sodium fluoride; Drug: Sodium monoflurophosphate; Drug: Sterile water
- Placebo Dentifrice + Sterile Water Rinse (Placebo Comparator): Placebo dentifrice and sterile water rinse
  Interventions: Drug: Sterile water

INTERVENTIONS:
Drug: Sodium fluoride — Test fluoride toothpaste and test fluoride mouth rinse
  Arms: Placebo Dentifrice + Test MR; Reference Dentifrice + Sterile Water Rinse; Test Dentifrice + Sterile Water Rinse; Test Dentifrice + Test Mouth Rinse (MR)
Drug: Sodium monoflurophosphate — United Kingdom marketed fluoride toothpaste
  Arms: Reference Dentifrice + Sterile Water Rinse
Drug: Sterile water — Sterile water rinse
  Arms: Placebo Dentifrice + Sterile Water Rinse; Reference Dentifrice + Sterile Water Rinse; Test Dentifrice + Sterile Water Rinse

SUMMARY:
An in situ model will be used to evaluate and compare enamel remineralization of bovine enamel specimens.

ELIGIBILITY:
Inclusion Criteria:

* An intact maxillary dental arch suitable for the retention of the palatal appliance and an intact mandibular dental arch - subjects may have fixed bridges replacing missing teeth
* No current active caries or periodontal disease that may compromise the study or the health of the subjects
* A gum base stimulated whole saliva flow rate greater than or equal to 0.8 mL/minute and an unstimulated whole saliva flow rate greater than or equal to 0.2 mL/minute

Exclusion Criteria:

* Known or suspected intolerance or hypersensitivity to the study materials (or closely related compounds) or any of their stated ingredients

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2009-08; Primary Completion 2009-10 (Actual); Study Completion 2009-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- Indiana University School of Dentistry, Indianapolis, Indiana, United States

REFERENCES:
- [Background] Maggio B, Guibert RG, Mason SC, Karwal R, Rees GD, Kelly S, Zero DT. Evaluation of mouthrinse and dentifrice regimens in an in situ erosion remineralisation model. J Dent. 2010 Nov;38 Suppl 3:S37-44. doi: 10.1016/S0300-5712(11)70007-0. PMID 21256403

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited at the clinical site.
Pre-assignment Details: Two days, prior to each treatment visit ,participants used a fluoride- free dentifrice twice daily to avoid any carry over effect.
Groups:
- Test Dentifrice + Test Mouth Rinse (MR): Participants were administered with treatment regimen comprising of test sodium fluoride (NaF) dentifrice [containing 1450 parts per million (ppm) fluoride (F) as NaF and potassium nitrate (KNO3)] and test NaF (450ppmF) MR. The treatment regimen included application of 1.5 gram (g) test NaF dentifrice to a wet study toothbrush, brushing for 25 seconds to create dentifrice slurry, swished the slurry around the mouth for one minute. After one minute, participants expectorated the slurry and rinsed the mouth with tap water. One hour later, the participants rinsed the mouth with 15mL of test MR for one minute.
- Test Dentifrice + Sterile Water Rinse: Participants were administered with treatment regimen comprising of test NaF Dentifrice (1450ppmF) and placebo sterile water rinse. The treatment regimen included application of 1.5g test NaF dentifrice to a wet study toothbrush, brushing for 25 seconds to create a dentifrice slurry, swished the slurry around the mouth for one minute. After one minute, participants expectorated the slurry and rinsed the mouth with tap water. One hour later, the participants rinsed the mouth with 15mL of sterile water rinse for one minute.
- Reference Dentifrice + Sterile Water Rinse: Participants were administered with treatment regimen comprising of reference sodium monofluorophosphate (NaMFP)/ NaF dentifrice (1450ppmF) and placebo sterile water MR. The treatment regimen included application of 1.5g reference dentifrice to a wet study toothbrush, brushing for 25 seconds to create a dentifrice slurry, swished the slurry around the mouth for one minute. After one minute, participants expectorated the slurry and rinsed the mouth with tap water. One hour later, the participants rinsed the mouth with 15mL of sterile water rinse for one minute.
- Placebo Dentifrice + Sterile Water Rinse: Participants were administered with treatment regimen comprising of placebo dentifrice (0ppmF) and placebo sterile water MR. The treatment regimen included application of 1.5g placebo dentifrice to a wet study toothbrush, brushing for 25 seconds to create a dentifrice slurry, swished the slurry around the mouth for one minute. After one minute, participants expectorated the slurry and rinsed the mouth with tap water. One hour later, the participants rinsed the mouth with 15mL of sterile water rinse for one minute.
- Placebo Dentifrice + Test MR: Participants were administered with treatment regimen comprising of placebo dentifrice (0ppmF) and test MR containing NaF (450ppmF). The treatment regimen included application of 1.5g placebo dentifrice to a wet study toothbrush, brushing for 25 seconds to create a dentifrice slurry, swished the slurry around the mouth for one minute. After one minute, participants expectorated the slurry and rinsed the mouth with tap water. One hour later, the participants rinsed the mouth with 15mL of test MR for one minute.
Period: Period I
Arm/Group | Test Dentifrice + Test Mouth Rinse (MR) | Test Dentifrice + Sterile Water Rinse | Reference Dentifrice + Sterile Water Rinse | Placebo Dentifrice + Sterile Water Rinse | Placebo Dentifrice + Test MR
Started | 7 | 7 | 7 | 7 | 8
Completed | 7 | 7 | 7 | 7 | 8
Not Completed | 0 | 0 | 0 | 0 | 0
Period: Period II
Arm/Group | Test Dentifrice + Test Mouth Rinse (MR) | Test Dentifrice + Sterile Water Rinse | Reference Dentifrice + Sterile Water Rinse | Placebo Dentifrice + Sterile Water Rinse | Placebo Dentifrice + Test MR
Started | 7 (Due to cross over design, different set of participants received this treatment compared to Period I) | 7 (Due to cross over design, different set of participants received this treatment compared to Period I) | 7 (Due to cross over design, different set of participants received this treatment compared to Period I) | 8 (Due to cross over design, different set of participants received this treatment compared to Period I) | 7 (Due to cross over design, different set of participants received this treatment compared to Period I)
Completed | 7 | 7 | 7 | 8 | 7
Not Completed | 0 | 0 | 0 | 0 | 0
Period: Period III
Arm/Group | Test Dentifrice + Test Mouth Rinse (MR) | Test Dentifrice + Sterile Water Rinse | Reference Dentifrice + Sterile Water Rinse | Placebo Dentifrice + Sterile Water Rinse | Placebo Dentifrice + Test MR
Started | 7 (Due to crossover design, different set of participants received this treatment compared to Period II) | 7 (Due to crossover design, different set of participants received this treatment compared to Period II) | 8 (Due to crossover design, different set of participants received this treatment compared to Period II) | 7 (Due to crossover design, different set of participants received this treatment compared to Period II) | 7 (Due to crossover design, different set of participants received this treatment compared to Period II)
Completed | 7 | 7 | 8 | 7 | 7
Not Completed | 0 | 0 | 0 | 0 | 0
Period: Period IV
Arm/Group | Test Dentifrice + Test Mouth Rinse (MR) | Test Dentifrice + Sterile Water Rinse | Reference Dentifrice + Sterile Water Rinse | Placebo Dentifrice + Sterile Water Rinse | Placebo Dentifrice + Test MR
Started | 7 (Due to crossover design,different set of participants received this treatment compared to Period III) | 8 (Due to crossover design,different set of participants received this treatment compared to Period III) | 7 (Due to crossover design,different set of participants received this treatment compared to Period III) | 7 (Due to crossover design,different set of participants received this treatment compared to Period III) | 7 (Due to crossover design,different set of participants received this treatment compared to Period III)
Completed | 7 | 8 | 7 | 7 | 7
Not Completed | 0 | 0 | 0 | 0 | 0
Period: Period V
Arm/Group | Test Dentifrice + Test Mouth Rinse (MR) | Test Dentifrice + Sterile Water Rinse | Reference Dentifrice + Sterile Water Rinse | Placebo Dentifrice + Sterile Water Rinse | Placebo Dentifrice + Test MR
Started | 8 (Due to crossover design, different set of participants received this treatment compared to Period IV) | 7 (Due to crossover design, different set of participants received this treatment compared to Period IV) | 7 (Due to crossover design, different set of participants received this treatment compared to Period IV) | 7 (Due to crossover design, different set of participants received this treatment compared to Period IV) | 7 (Due to crossover design, different set of participants received this treatment compared to Period IV)
Completed | 8 | 7 | 7 | 7 | 7
Not Completed | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- All Study Participants: All randomized participants were included for baseline evaluation.
Arm/Group | All Study Participants
Number analyzed (Participants) | 36
Age, Continuous [Mean (Standard Deviation); unit: Years] | 37.0 (12.90)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19
  Male | 17
Region of Enrollment [Number; unit: Participants]
  United States | 36

OUTCOME MEASURES:

1. Primary Outcome: Adjusted Mean Percent Net Erosion Resistance (NER) of Enamel Specimens Exposed to Test Dentifrice + Test MR Relative to: 1) Test Dentifrice+ Sterile Water Rinse 2) Reference Dentifrice+ Sterile Water Rinse 3) Placebo Dentifrice+ Sterile Water Rinse
Description: Enamel specimens were exposed to dietary erosive challenge and set of five indentations within each specimen was measured. Decrease in the indentation length compared to the baseline indicates hardening of enamel surface. Enamel specimens were exposed to second erosion challenge to determine NER which compared the indentations values of enamel specimens at baseline (B), first erosive (E1) and second erosive challenge (E2). Percent NER was calculated by formula: [(E1-E2)/ (E1-B)]*100. Smaller the negative NER, better is treatment regimen in imparting resistance to enamel.
Time Frame: Baseline, 4 hours post treatment in each treatment period
Population: Per protocol (PP) population: All randomized subjects who received at least one dose of the study treatments and had no major protocol deviations were included in analysis.
Measure: Least Squares Mean (Standard Error); unit: Percent NER
Groups:
- Test Dentifrice + Test MR: Participants were administered with treatment regimen comprising of test NaF dentifrice [containing 1450ppmF as NaF and KNO3] and test NaF (450ppmF) MR. The treatment regimen included application of 1.5g test NaF dentifrice to a wet study toothbrush, brushing for 25 seconds to create a dentifrice slurry, swished the slurry around the mouth for one minute. After one minute, participants expectorated the slurry and rinsed the mouth with tap water. One hour later, the participants rinsed the mouth with 15mL of test MR for one minute.
- Test Dentifrice + Sterile Water Rinse: Participants were administered with treatment regimen comprising of test NaF Dentifrice (1450ppmF) and placebo sterile water rinse. The treatment regimen included application of 1.5g test NaF dentifrice to a wet study toothbrush, brushing for 25 seconds to create dentifrice slurry, swished the slurry around the mouth for one minute. After one minute, participants expectorated the slurry and rinsed the mouth with tap water. One hour later, the participants rinsed the mouth with 15mL of sterile water rinse for one minute.
- Reference Dentifrice + Sterile Water Rinse: Participants were administered with treatment regimen comprising of reference NaMFP/ NaF dentifrice (1450ppmF) and placebo sterile water MR. The treatment regimen included application of 1.5g reference dentifrice to a wet study toothbrush, brushing for 25 seconds to create dentifrice slurry, swished the slurry around the mouth for one minute. After one minute, participants expectorated the slurry and rinsed the mouth with tap water. One hour later, the participants rinsed the mouth with 15mL of sterile water rinse for one minute.
- Placebo Dentifrice + Sterile Water Rinse: Participants were administered with treatment regimen comprising of placebo dentifrice (0ppmF) and placebo sterile water MR. The treatment regimen included application of 1.5g placebo dentifrice to a wet study toothbrush, brushing for 25 seconds to create dentifrice slurry, swished the slurry around the mouth for one minute. After one minute, participants expectorated the slurry and rinsed the mouth with tap water. One hour later, the participants rinsed the mouth with 15mL of sterile water rinse for one minute.
Arm/Group | Test Dentifrice + Test MR | Test Dentifrice + Sterile Water Rinse | Reference Dentifrice + Sterile Water Rinse | Placebo Dentifrice + Sterile Water Rinse
Number analyzed (Participants) | 36 | 36 | 36 | 36
Percent NER | -2.88 (2.155) | -14.54 (2.155) | -29.48 (2.155) | -40.05 (2.155)
Statistical Analysis 1: Comparison: Test Dentifrice + Test MR vs Test Dentifrice + Sterile Water Rinse; Null hypothesis considered population means for the test dentifrice+ test MR treatment regimen and test dentifrice + sterile water rinse treatment regimen to be equal with respect to percent NER. Statistical tests were 2-sided with a significance level of 0.05; Test type: Superiority or Other; p < 0.0001, ANOVA — No adjustments made for multiple comparisons as the primary comparison was pre-specified; ANOVA with factors for treatment, study period, and subject (random effect); Adjusted Mean Difference = 11.66, 95% CI 2-sided [7.09 to 16.24] — Difference is first named treatment minus second named treatment such that a positive difference favours the first named treatment
Statistical Analysis 2: Comparison: Test Dentifrice + Test MR vs Reference Dentifrice + Sterile Water Rinse; Null hypothesis considered population means for the test dentifrice+ test MR treatment regimen and reference dentifrice + sterile water rinse treatment regimen to be equal with respect to percent NER. Statistical tests were 2-sided with a significance level of 0.05; Test type: Superiority or Other; p < 0.0001, ANOVA — No adjustments made for multiple comparisons as primary comparison was pre-specified; ANOVA with factors for treatment, study period, and subject (random effect); Adjusted Mean DIfference = 26.6, 95% CI 2-sided [22.02 to 31.18] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: Test Dentifrice + Test MR vs Placebo Dentifrice + Sterile Water Rinse; Null hypothesis considered population means for the test dentifrice+ test MR treatment regimen and placebo dentifrice + sterile water rinse treatment regimen to be equal with respect to percent NER. Statistical tests were 2-sided with a significance level of 0.05; Test type: Superiority or Other; p < 0.0001, ANOVA — No adjustments made for multiple comparisons as the primary comparison was pre-specified; ANOVA with factors for treatment, study period, and subject (random effect); Adjusted Mean Difference = 37.17, 95% CI 2-sided [32.59 to 41.74] — [estimate comment as in outcome 1, analysis 1]

2. Secondary Outcome: Adjusted Mean Percentage Surface Microhardness (SMH) Recovery of Enamel Specimens Exposed to Test Dentifrice + Test MR Relative to: 1)Test Dentifrice+Sterile Water Rinse 2)Reference Dentifrice+Sterile Water Rinse 3)Placebo Dentifrice+ Sterile Water Rinse
Description: SMH test was used to assess mineralization status of enamel specimens using a Wilson 2100 Hardness tester. SMH was determined by measuring the length of the indentations of enamel specimens. An increase in the indentation length compared to the baseline indicates softening while decrease in the indentation length represents rehardening of enamel surface. Percent SMH recovery was calculated from indentation values of enamel specimens at baseline (B), after in-situ hardening (R) and after first erosive challenge (E1) using formula: [(E1-R)/ (E1-B)]*100.
Time Frame: Baseline, 4 hours post treatment in each treatment period.
Population: PP population: All randomized participants who received at least one dose of the study treatments and had no major protocol deviations were included in analysis.
Measure: Least Squares Mean (Standard Error); unit: Percent SMH
Arm/Group | Test Dentifrice + Test MR | Test Dentifrice + Sterile Water Rinse | Reference Dentifrice + Sterile Water Rinse | Placebo Dentifrice + Sterile Water Rinse
Number analyzed (Participants) | 36 | 36 | 36 | 36
Percent SMH | 42.14 (1.399) | 38.02 (1.399) | 30.88 (1.399) | 30.57 (1.399)
Statistical Analysis 1: Comparison: Test Dentifrice + Test MR vs Test Dentifrice + Sterile Water Rinse; Null hypothesis considered population means for the test dentifrice+ test MR treatment regimen and test dentifrice + Sterile water rinse to be equal with respect to percent SMH recovery. Statistical tests were 2-sided with a significance level of 0.05; Test type: Superiority or Other; p = 0.0083, ANOVA — No adjustments made for multiple comparisons as the primary comparison was pre-specified; ANOVA with factors for treatment, study period, and subject (random effect); Adjusted Mean Difference = 4.11, 95% CI 2-sided [1.07 to 7.15] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Test Dentifrice + Test MR vs Reference Dentifrice + Sterile Water Rinse; Null hypothesis considered population means for the test dentifrice+ test MR treatment regimen and reference dentifrice + Sterile water rinse treatment regimen to be equal with respect to percent SMH recovery. Statistical tests were 2-sided with a significance level of 0.05; Test type: Superiority or Other; p < 0.0001, ANOVA — No adjustments made for multiple comparisons as the primary comparison was pre-specified; ANOVA with factors for treatment, study period, and subject (random effect); Adjusted Mean DIfference = 11.25, 95% CI 2-sided [8.22 to 14.29] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: Test Dentifrice + Test MR vs Placebo Dentifrice + Sterile Water Rinse; Null hypothesis considered population means for the test dentifrice+ test MR treatment regimen and placebo dentifrice + Sterile water rinse treatment regimen to be equal with respect to percent SMH recovery. Statistical tests were 2-sided with a significance level of 0.05; Test type: Superiority or Other; p < 0.0001, ANOVA — No adjustments made for multiple comparisons as the primary comparison was pre-specified; ANOVA with factors for treatment, study period, and subject (random effect); Adjusted Mean Difference = 11.56, 95% CI 2-sided [8.53 to 14.60] — [estimate comment as in outcome 1, analysis 1]

3. Other Pre Specified Outcome: Adjusted Mean Percent NER of Enamel Specimens Exposed to a Treatment Regimen of Placebo Dentifrice + Test MR Relative to: 1) Test Dentifrice +Test MR 2) Test Dentifrice + Sterile Water Rinse 3) Reference Dentifrice +Sterile Water Rinse
Description: as for outcome 1
Time Frame: Baseline, 4 hours post treatment in each treatment period
Population: PP population: All randomized subjects who received at least one dose of the study treatments and had no major protocol deviations were included in analysis.
Measure: Least Squares Mean (Standard Error); unit: Percent NER
Arm/Group | Placebo Dentifrice + Test MR | Test Dentifrice + Test MR | Test Dentifrice + Sterile Water Rinse | Reference Dentifrice + Sterile Water Rinse | Placebo Dentifrice + Sterile Water Rinse
Number analyzed (Participants) | 36 | 36 | 36 | 36 | 36
Percent NER | -3.76 (2.155) | -2.88 (2.155) | -14.54 (2.155) | -29.48 (2.155) | -40.05 (2.155)
Statistical Analysis 1: Comparison: Placebo Dentifrice + Test MR vs Test Dentifrice + Test MR; Null hypothesis considered population means for the Placebo Dentifrice + Test MR and Test dentifrice+ Test MR treatment regimen treatment regimen to be equal with respect to percent NER. Statistical tests were 2-sided with a significance level of 0.05; Test type: Superiority or Other; p = 0.7041, ANOVA — No adjustments made for multiple comparisons as the primary comparison was pre-specified; ANOVA with factors for treatment, study period, and subject (random effect); Adjusted Mean Difference = -0.88, 95% CI 2-sided [-5.46 to 3.69] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Placebo Dentifrice + Test MR vs Test Dentifrice + Sterile Water Rinse; Null hypothesis considered population means for the Placebo dentifrice+ test MR treatment regimen and test dentifrice + sterile water rinse treatment regimen to be equal with respect to percent NER. Statistical tests were 2-sided with a significance level of 0.05; Test type: Superiority or Other; p < 0.0001, ANOVA — No adjustments made for multiple comparisons as the primary comparison was pre-specified; ANOVA with factors for treatment, study period, and subject (random effect); Adjusted Mean Difference = 10.78, 95% CI 2-sided [6.21 to 15.36] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: Placebo Dentifrice + Test MR vs Reference Dentifrice + Sterile Water Rinse; Null hypothesis considered population means for the Placebo dentifrice+ Test MR treatment regimen and Reference dentifrice + sterile water rinse treatment regimen to be equal with respect to percent NER. Statistical tests were 2-sided with a significance level of 0.05; Test type: Superiority or Other; p < 0.0001, ANOVA — No adjustments made for multiple comparisons as the primary comparison was pre-specified; ANOVA with factors for treatment, study period, and subject (random effect); Adjusted Mean Difference = 25.72, 95% CI 2-sided [21.14 to 30.29] — Difference is first named treatment minus second named treatment such that a positive difference favors the first named treatment
Statistical Analysis 4: Comparison: Placebo Dentifrice + Test MR vs Placebo Dentifrice + Sterile Water Rinse; Null hypothesis considered population means for the Placebo dentifrice+ test MR treatment regimen and Placebo dentifrice + sterile water rinse treatment regimen to be equal with respect to percent NER. Statistical tests were 2-sided with a significance level of 0.05; Test type: Superiority or Other; p < 0.0001, ANOVA — No adjustments made for multiple comparisons as the primary comparison was pre-specified; ANOVA with factors for treatment, study period, and subject (random effect); Adjusted Mean Difference = 36.29, 95% CI 2-sided [31.71 to 40.86] — [estimate comment as in outcome 1, analysis 1]

4. Other Pre Specified Outcome: Adjusted Mean Percentage SMH Recovery of Enamel Specimens Exposed to Test Dentifrice + Test MR Relative to Following Treatment Regimens: 1) Test Dentifrice +Test MR 2) Test Dentifrice + Sterile Water 3) Reference Dentifrice +Sterile Water
Description: as for outcome 2
Time Frame: Baseline, 4 hours post treatment in each treatment period
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: Percent SMH
Arm/Group | Placebo Dentifrice + Test MR | Test Dentifrice + Test MR | Test Dentifrice + Sterile Water Rinse | Reference Dentifrice + Sterile Water Rinse | Placebo Dentifrice + Sterile Water Rinse
Number analyzed (Participants) | 36 | 36 | 36 | 36 | 36
Percent SMH | 37.75 (1.399) | 42.14 (1.399) | 38.02 (1.399) | 30.88 (1.399) | 30.57 (1.399)
Statistical Analysis 1: Comparison: Placebo Dentifrice + Test MR vs Test Dentifrice + Test MR; Null hypothesis considered population means for the Placebo dentifrice+ Test MR treatment regimen and Test dentifrice + Test MR to be equal with respect to percent SMH recovery. Statistical tests were 2-sided with a significance level of 0.05; Test type: Superiority or Other; p = 0.0049, ANOVA — No adjustments made for multiple comparisons as the primary comparison was pre-specified; ANOVA with factors for treatment, study period, and subject (random effect); Adjusted Mean Difference = -4.39, 95% CI 2-sided [-7.43 to -1.35] — [estimate comment as in outcome 3, analysis 3]
Statistical Analysis 2: Comparison: Placebo Dentifrice + Test MR vs Test Dentifrice + Sterile Water Rinse; Null hypothesis considered population means for the Placebo dentifrice+ test MR treatment regimen and test dentifrice + sterile water rinse to be equal with respect to percent SMH recovery. Statistical tests were 2-sided with a significance level of 0.05; Test type: Superiority or Other; p = 0.8571, ANOVA — No adjustments made for multiple comparisons as the primary comparison was pre-specified; ANOVA with factors for treatment, study period, and subject (random effect); Adjusted Mean Difference = -0.28, 95% CI 2-sided [-3.31 to 2.76] — [estimate comment as in outcome 3, analysis 3]
Statistical Analysis 3: Comparison: Placebo Dentifrice + Test MR vs Reference Dentifrice + Sterile Water Rinse; Null hypothesis considered population means for the Placebo Dentifrice + Test MR treatment regimen and Reference Dentifrice + Sterile water rinse to be equal with respect to percent SMH recovery. Statistical tests were 2-sided with a significance level of 0.05; Test type: Superiority or Other; p < 0.0001, ANOVA — No adjustments made for multiple comparisons as the primary comparison was pre-specified; ANOVA with factors for treatment, study period, and subject (random effect); Adjusted Mean Difference = 6.87, 95% CI 2-sided [3.83 to 9.90] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 4: Comparison: Placebo Dentifrice + Test MR vs Placebo Dentifrice + Sterile Water Rinse; Null hypothesis considered population means for the Placebo Dentifrice + Test MR treatment regimen and Placebo dentifrice + Sterile water rinse to be equal with respect to percent SMH recovery. Statistical tests were 2-sided with a significance level of 0.05; Test type: Superiority or Other; p < 0.0001, ANOVA — No adjustments made for multiple comparisons as the primary comparison was pre-specified; ANOVA with factors for treatment, study period, and subject (random effect); Adjusted Mean Difference = 7.17, 95% CI 2-sided [4.14 to 10.21] — [estimate comment as in outcome 3, analysis 3]

5. Other Pre Specified Outcome: Adjusted Mean Percent NER of Enamel Specimens Exposed to Test Dentifrice +Sterile Water Rinse and Reference Dentifrice +Sterile Water Rinse
Description: as for outcome 1
Time Frame: Baseline, 4 hours post treatment in each treatment period
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: Percent NER
Arm/Group | Test Dentifrice + Sterile Water Rinse | Reference Dentifrice + Sterile Water Rinse
Number analyzed (Participants) | 36 | 36
Percent NER | -2.88 (2.155) | -29.48 (2.155)
Statistical Analysis 1: Comparison: Test Dentifrice + Sterile Water Rinse vs Reference Dentifrice + Sterile Water Rinse; Null hypothesis considered population means for the Test Dentifrice + Sterile water rinse treatment regimen andReference Dentifrice + Sterile water rinse treatment regimen to be equal with respect to percent NER. Statistical tests were 2-sided with a significance level of 0.05; Test type: Superiority or Other; ANOVA — No adjustments made for multiple comparisons as the primary comparison was pre-specified; ANOVA with factors for treatment, study period, and subject (random effect); Adjusted Mean Difference = 14.94, 95% CI 2-sided [10.36 to 19.51] — [estimate comment as in outcome 1, analysis 1]

6. Other Pre Specified Outcome: Adjusted Mean Percent SMH Recovery of Enamel Specimens Exposed to Test Dentifrice +Sterile Water Rinse and Reference Dentifrice +Sterile Water Rinse
Description: as for outcome 2
Time Frame: Baseline, 4 hours post treatment in each treatment period
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: Percent SMH
Arm/Group | Test Dentifrice + Sterile Water Rinse | Reference Dentifrice + Sterile Water Rinse
Number analyzed (Participants) | 36 | 36
Percent SMH | 38.02 (1.399) | 30.88 (1.399)
Statistical Analysis 1: Comparison: Test Dentifrice + Sterile Water Rinse vs Reference Dentifrice + Sterile Water Rinse; Null hypothesis considered population means for the Test Dentifrice + Sterile water rinse treatment regimen and Reference Dentifrice + Sterile water rinse to be equal with respect to percent SMH recovery. Statistical tests were 2-sided with a significance level of 0.05; Test type: Superiority or Other; p < 0.0001, ANOVA — No adjustments made for multiple comparisons as the primary comparison was pre-specified; ANOVA with factors for treatment, study period, and subject (random effect); Adjusted Mean Difference = 7.14, 95% CI 2-sided [4.11 to 10.18] — [estimate comment as in outcome 1, analysis 1]

ADVERSE EVENTS:
Time Frame: All AEs encountered or spontaneously reported following administration of any investigational product (including washout product), or for up to 5 days after the last administration of investigational product were recorded.
Groups:
- Placebo Dentifrice + Test MR: Participants were administered with treatment regimen comprising of placebo dentifrice (0ppmF) and test MR containing NaF (450ppmF). The treatment regimen included application of 1.5g placebo dentifrice to a wet study toothbrush, brushing for 25 seconds to create dentifrice slurry, swished the slurry around the mouth for one minute. After one minute, participants expectorated the slurry and rinsed the mouth with tap water. One hour later, the participants rinsed the mouth with 15mL of test MR for one minute.
Arm/Group | Test Dentifrice + Test MR | Test Dentifrice + Sterile Water Rinse | Reference Dentifrice + Sterile Water Rinse | Placebo Dentifrice + Test MR | Placebo Dentifrice + Sterile Water Rinse
Serious Adverse Events (participants affected / at risk) | 0/36 | 0/36 | 0/36 | 0/36 | 0/36
Other Adverse Events (participants affected / at risk) | 0/36 | 1/36 | 2/36 | 1/36 | 0/36
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Test Dentifrice + Test MR (N=36) | Test Dentifrice + Sterile Water Rinse (N=36) | Reference Dentifrice + Sterile Water Rinse (N=36) | Placebo Dentifrice + Test MR (N=36) | Placebo Dentifrice + Sterile Water Rinse (N=36)
Gingival Erythema (Gastrointestinal disorders) | 0 (0) | 1 (1) | 2 (2) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.